CLINICAL TRIAL: NCT06163807
Title: Follow-up of Spanish Prospective Asthma and Nasal Polyposis Registry
Acronym: MEGA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: SGZ-2022-13739
Record Dates: First submitted 2023-11-02; First posted 2023-12-11 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-10

CONDITIONS: Chronic Asthma
Keywords: asthma; biologics; biomarkers; nasal polyposis; eosinophils
MeSH Terms: conditions — Asthma; Nasal Polyps | interventions — Anti-Asthmatic Agents; Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood cells, sputum cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asthma patients with different severities: Asthma patients with different severities followed for 5 years. Real-life, antiasthmatic drugs selected by investigators. Clinical, analytical, biomarkers, image techniques
  Interventions: Drug: Antiasthmatic
- Severe asthma patients treated with biologics: In follow-up for 3 years and new patients. Real-life, antiasthmatic drugs selected by investigators. Clinical, analytical, biomarkers, image techniques
  Interventions: Drug: Antiasthmatic

INTERVENTIONS:
Drug: Antiasthmatic — real-life
  Other Names: biologics

SUMMARY:
Primary objective

- To study the stability of different phenotypes and endotypes of asthma at 3, 5, and 7 years of follow-up and - in MEGA COHORT and in patients on biologic treatment

Secondary objective(s)

* To study biomarkers variation post-treatment in patients with and without Nasal Polyposis
* To demonstrate the existence of different subtypes of eosinophils that may be phenotypically and functionally heterogeneous
* To increase the number of patients in the cohort on biologic treatment to reach at least 900 (400 over the current cohort).

DETAILED DESCRIPTION:
Open-labeled National, Multicenter Non-interventional on the therapeutic strategy, Prospective (longitudinal) Disease registry, 3 years of follow-up

1. Correlation between non-invasive T2 markers (FeNO, blood eosinophils) versus inflammatory markers in sputum (eosinophils, periostin, NO, etc.)
2. Cluster analysis in both cohorts.
3. Analysis of some treatable traits on asthma control in MEGA cohort (BMI, anxiety and depression scale, exercise).
4. To characterize exacerbations (numbers, ICU admissions, treatments compliance, etc).
5. Analysis of compliance with asthma medications.
6. Analysis of patients with phenotype T2-LOW in MEGA cohort.
7. Analysis of patients with undetectable total IgE ( < 10 UI/L).
8. Role of microRNA in diagnosis, follow-up and variations after treatments.
9. Analysis of alarmins (TSLP, IL-33 e IL-25) and IL-6 in blood and sputum.
10. To Immunophenotype eosinophils by single-cell analysis in blood and sputum at baseline and post-biological treatment.

ELIGIBILITY:
Inclusion Criteria:

For the general asthma cohort (MEGA):

* Age from 18 to 80 y.o. with asthma with and without nasal polyposis based on GINA guidelines (compatible clinical symptoms+reversibility of at least 12% and 200 mL in FEV1 after the administration of 200-400 μg albuterol/salbutamol or positive methacholine test) of several severities attended at participant centres
* Already in follow-up in MEGA cohort
* To participate in the study
* Signed informed consent

Inclusion criteria for asthma patients treated with biologics

* Patients from 18 to 80 y.o. with uncontrolled asthma with and without nasal polyposis that fulfil criteria to be treated with biological drugs (Existing treatment with medium-to-high-dose ICS (≥ 250 μg of fluticasone propionate twice daily or equipotent ICS daily dosage to a maximum of 2000 μg/day of fluticasone propionate or equivalent) in combination with a second controller (e.g., LABA, LTRA) for at least 3 months+ airflow limitation- FEV1 <80%/FEV1/FVC <70+ACQ-5 score ≥ 1.5/ ACT < 19 at inclusion and/or have experience any of the following events on the last year: treatment with systemic steroids/ hospitalization or emergency medical care visit for worsening asthma.
* When planning dupilumab, mepolizumab, benralizumab or reslizumab, biomarker levels, and exacerbation in the previous year will be considered according to the Spanish Ministry of Health recommendations for reimbursement of any biological drug in severe asthma. In the case of Omalizumab allergic asthma and IgE > 75 and < 1500 UI
* Patients already in follow-up in the cohort of patients treated with biologics
* Willing to participate in the study
* Sign informed consent

Exclusion Criteria:

* Exclusion criteria for MEGA COHORT

  * Diagnosis of chronic obstructive pulmonary disease or other lung disease that may impair lung function
  * Comorbid disease that might interfere with the evaluation, e.g. psychiatric disorders
  * Patients participating in other clinical trials
  * Patients without the capacity to understand the aim of the study
* Exclusion criteria for asthma patients treated with biologics

  * Diagnosis of chronic obstructive pulmonary disease or other lung disease that may impair lung function
  * Comorbid disease that might interfere with the evaluation, e.g. psychiatric disorders
  * Patients participating in other clinical trials
  * Patients without the capacity to understand the aim of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with asthma (intermittent, mild, moderate or severe asthma according to the GINA classification), with or without nasal polyposis attended third-level hospitals of the Spanish National Health System.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between non-invasive T2 biomarkers versus biomarkers in sputum | at date of randomization and after one year of follow-up
  biomarkers in blood (eosinophils, mRNA, periostine), exhaled nitric oxide (FeNO), sputum cell analysis and mRNA expression

SECONDARY OUTCOMES:
Analysis of treatable traits on asthma control by ACT questionnaire | at date of randomization and after one, two and three years of follow-up
  asthma control by Asthma Control Questionnaire (ACT)
To characterize asthma exacerbations. | at date of randomization and after one, two and three years of follow-up
  number of exacerbations, type of exacerbation, ICU admissions, treatment compliance
Analysis of withdrawing asthma medications | at date of randomization and after one, two and three years of follow-up
  percentage of anti-asthmatic medication withdrawn from the pharmacy in the electronic prescription with respect to that prescribed in your treatment
Analysis of patients with phenotype T2-LOW (IgE less than 75 kU/L, blood eosinophils less than 150 cells/μL, and FeNO less than 20 ppb) | at date of randomization and after one year of follow-up
  number of exacerbations
Analysis of clinical outcomes, pulmonary function tests, biomarkers patients with very low total IgE ( < 10 UI/L) | at date of randomization and after one year of follow-up
  Total IgE
Role of alarmins and IL-6 in the component of inflammation in asthma | at date of randomization and after one year of follow-up
  measure of TSLP, IL-33 e IL-25 in blood and sputum
Role of microRNAs in asthma diagnosis and variations after different treatments | 1 year
  expression of mRNAs in blood and sputum
Immunophenotype eosinophils | 1 year
  single-cell analysis of eosinophils in blood and sputum at baseline
Stability of asthma phenotypes along the follow-up | at date of randomization and after one, two and three years of follow-up
  % of eosinophils in sputum sample

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Sastre, Study Director — Fundacion Jimenez Diaz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dominguez-Ortega J, Luna-Porta JA, Olaguibel JM, Barranco P, Arismendi E, Barroso B, Betancor D, Bobolea I, Caballero ML, Cardaba B, Cruz MJ, Curto E, Gonzalez-Barcala FJ, Losantos-Garcia I, Martinez-Rivera C, Mendez-Brea P, Mullol J, Munoz X, Picado C, Plaza V, Del Pozo V, Rial MJ, Sastre J, Soto L, Valero A, Valverde-Monge M, Quirce S. Exacerbations Among Patients With Asthma Are Largely Dependent on the Presence of Multimorbidity. J Investig Allergol Clin Immunol. 2023 Jul 27;33(4):281-288. doi: 10.18176/jiaci.0816. Epub 2002 May 3. PMID 35503227
- [Result] Matabuena M, Salgado FJ, Nieto-Fontarigo JJ, Alvarez-Puebla MJ, Arismendi E, Barranco P, Bobolea I, Caballero ML, Canas JA, Cardaba B, Cruz MJ, Curto E, Dominguez-Ortega J, Luna JA, Martinez-Rivera C, Mullol J, Munoz X, Rodriguez-Garcia J, Olaguibel JM, Picado C, Plaza V, Quirce S, Rial MJ, Romero-Mesones C, Sastre B, Soto-Retes L, Valero A, Valverde-Monge M, Del Pozo V, Sastre J, Gonzalez-Barcala FJ. Identification of Asthma Phenotypes in the Spanish MEGA Cohort Study Using Cluster Analysis. Arch Bronconeumol. 2023 Apr;59(4):223-231. doi: 10.1016/j.arbres.2023.01.007. Epub 2023 Jan 18. English, Spanish. PMID 36732158
- [Result] Rodrigo-Munoz JM, Canas JA, Sastre B, Rego N, Greif G, Rial M, Minguez P, Mahillo-Fernandez I, Fernandez-Nieto M, Mora I, Barranco P, Quirce S, Sastre J, Del Pozo V. Asthma diagnosis using integrated analysis of eosinophil microRNAs. Allergy. 2019 Mar;74(3):507-517. doi: 10.1111/all.13570. Epub 2018 Oct 11. PMID 30040124
- [Result] Romero-Mesones C, Cruz MJ, Alobid I, Barroso B, Arismendi E, Barranco P, Betancor D, Bobolea I, Cardaba B, Curto E, Domenech G, Dominguez-Ortega J, Espejo D, Gonzalez-Barcala FJ, Luna-Porta JA, Martinez-Rivera C, Mendez-Brea P, Mullol J, Olaguibel JM, Picado C, Plaza V, Del Pozo V, Quirce S, Rial MJ, Rodrigo-Munoz JM, Sastre J, Serrano S, Soto-Retes L, Valero A, Valverde-Monge M, Munoz X. Disposition of Work-Related Asthma in a Spanish Asthma Cohort: Comparison of Asthma Severity Between Employed and Retired Workers. J Allergy Clin Immunol Pract. 2023 Nov;11(11):3407-3413.e1. doi: 10.1016/j.jaip.2023.06.040. Epub 2023 Jun 28. PMID 37391017
- [Result] Barroso B, Valverde-Monge M, Betancor D, Gomez-Lopez A, Villalobos-Vilda C, Gonzalez-Cano B, Sastre J. Improvement in Smell Using Monoclonal Antibodies Among Patients With Chronic Rhinosinusitis With Nasal Polyps: A Systematic Review. J Investig Allergol Clin Immunol. 2023 Dec 14;33(6):419-430. doi: 10.18176/jiaci.0939. Epub 2023 Sep 4. PMID 37669083
- [Result] Baos S, Calzada D, Cremades-Jimeno L, de Pedro M, Sastre J, Picado C, Quiralte J, Florido F, Lahoz C, Cardaba B. Discriminatory Molecular Biomarkers of Allergic and Nonallergic Asthma and Its Severity. Front Immunol. 2019 May 9;10:1051. doi: 10.3389/fimmu.2019.01051. eCollection 2019. PMID 31143187
- [Result] Baptista-Serna L, Rodrigo-Munoz JM, Minguez P, Valverde-Monge M, Arismendi E, Barranco P, Barroso B, Bobolea I, Canas JA, Cardaba B, Cruz MJ, Curto E, Dominguez-Ortega J, Garcia-Latorre R, Gonzalez-Barcala FJ, Martinez-Rivera C, Mullol J, Munoz X, Olaguibel JM, Picado C, Plaza V, Quirce S, Rial MJ, Sastre B, Soto L, Valero A, Del Pozo V, Sastre J. Anxiety and body mass index affect asthma control: data from a prospective Spanish cohort. J Allergy Clin Immunol Pract. 2022 Mar;10(3):863-866.e1. doi: 10.1016/j.jaip.2021.10.013. Epub 2021 Oct 18. No abstract available. PMID 34673289
- [Result] Rial MJ, Alvarez-Puebla MJ, Arismendi E, Caballero ML, Canas JA, Cruz MJ, Gonzalez-Barcala FJ, Luna JA, Martinez-Rivera C, Mullol J, Munoz X, Olaguibel JM, Picado C, Plaza V, Quirce S, Romero-Mesones C, Salgado FJ, Sastre B, Soto-Retes L, Valero A, Valverde M, Sastre J, Pozo VD. Clinical and inflammatory characteristics of patients with asthma in the Spanish MEGA project cohort. Clin Transl Allergy. 2021 Mar;11(1):e12001. doi: 10.1002/clt2.12001. PMID 33900052
- [Result] Betancor D, Olaguibel JM, Rodrigo-Munoz JM, Arismendi E, Barranco P, Barroso B, Bobolea I, Cardaba B, Cruz MJ, Curto E, Del Pozo V, Gonzalez-Barcala FJ, Martinez-Rivera C, Mullol J, Munoz X, Picado C, Plaza V, Quirce S, Rial MJ, Soto L, Valero A, Valverde-Monge M, Sastre J. How reliably can algorithms identify eosinophilic asthma phenotypes using non-invasive biomarkers? Clin Transl Allergy. 2022 Aug 20;12(8):e12182. doi: 10.1002/clt2.12182. eCollection 2022 Aug. PMID 36000018
- [Result] Rial MJ, Valverde M, Del Pozo V, Gonzalez-Barcala FJ, Martinez-Rivera C, Munoz X, Olaguibel JM, Plaza V, Curto E, Quirce S, Barranco P, Dominguez-Ortega J, Mullol J, Picado C, Valero A, Bobolea I, Arismendi E, Ribo P, Sastre J. Clinical characteristics in 545 patients with severe asthma on biological treatment during the COVID-19 outbreak. J Allergy Clin Immunol Pract. 2021 Jan;9(1):487-489.e1. doi: 10.1016/j.jaip.2020.09.050. Epub 2020 Oct 9. No abstract available. PMID 33045398